CLINICAL TRIAL: NCT02626507
Title: Phase I Dose-Escalation Study of Combination of Gedatolisib (a Dual Inhibitor of PI3-K and mTOR) With Palbociclib and Faslodex in the Neoadjuvant Setting in Previously Untreated Patients With ER+/HER2- Breast Cancer
Brief Title: Phase I Study of Combination of Gedatolisib With Palbociclib and Faslodex in Patients With ER+/HER2- Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hoffman Oncology (Other)
Collaborators: DSCS CRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL- Gedatolisib-001
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: ER+/HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — gedatolisib; Fulvestrant; palbociclib; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gedatolisib ER+/HER2- Breast Cancer (Experimental): * Gedatolisib at escalating doses of 180, 215 and 260 mg via a 3-6 dose-escalation scheme is administered once weekly on the first day for each of the four weeks during the four 4-week cycles.
  * Faslodex at 500 mg is administered IM into the buttocks slowly (over 1 - 2 minutes per injection) as two 5-mL injections, one in each buttock, on Days 1 and 15 of Cycle 1 and on Day 1 of the remaining three 4-week treatment cycles.
  * Palbociclib at 125 mg is administered PO with food daily on Days 1-21 for each of the four 4-week cycles
  * Zoladex is used to render menopause in pre-menopausal subjects, given once every 28 days starting at least 14 days prior to treatment.
  Interventions: Drug: Gedatolisib; Drug: Faslodex; Drug: Palbociclib; Drug: Zoladex

INTERVENTIONS:
Drug: Gedatolisib — adenosine triphosphate (ATP) competitive, highly selective and potent inhibitor of pan-class I isoform phosphatidylinositol-4,5-bisphosphate 3-kinase (PI3-K)
  Other Names: Code name PF-05212384; PKI-587
Drug: Faslodex — Faslodex® (Fulvestrant) is a potent anti-estrogen drug that binds and degrades estrogen receptors (ERs).
  Other Names: Fulvestrant
Drug: Palbociclib — Palbociclib (Ibrance®) is an orally active highly selective reversible inhibitor of cyclin-dependent kinase (CDK) 4 and CDK 6.
  Other Names: Ibrance
Drug: Zoladex — Zoladex is used to render menopause in pre-menopausal subjects, given once every 28 days starting at least 14 days prior to treatment.
  Other Names: goserelin

SUMMARY:
This is a dose-escalation Phase Ib clinical trial in 18 patients with newly diagnosed Stage I-IV ER+/HER2- breast cancer, with the primary cancer in place. These patients have not received prior therapy for their breast cancer and intend to undergo surgery after four cycles of therapy.

This is an open-label study, and investigators and subjects are not blinded to the treatment. The reason for using an open-label study design is because this is a dose-escalation trial, and the investigators need to determine the potential toxicity before a decision can be made to continue the dose escalation procedures.

The assignment of patients will not be randomized, as this is a dose-escalation trial.

DETAILED DESCRIPTION:
Palbociclib (Ibrance®) is an orally active highly selective reversible inhibitor of cyclin-dependent kinase (CDK) 4 and CDK 6. Faslodex® (Fulvestrant) is a potent anti-estrogen drug that binds and degrades estrogen receptors (ERs). Interim results from the Phase 3 trial (Study PALOMA-3) have shown that combination of palbociclib and Faslodex increases progressive-free survival (PFS) from 3.8 to 9.2 months in patients with metastatic estrogen receptor positive (ER+) and human epidermal growth factor receptor 2 negative (HER2-) breast cancer that progressed during or after anti-endocrine therapy (Turner et al. 2015). The palbociclib/Faslodex combination was found to be well tolerated. Additionally, there is growing data indicating that this combination can be safely and effectively administered up front in anti-endocrine therapy-naive patients in the neoadjuvant setting.

Gedatolisib (code name PF-05212384, formerly known as PKI-587) is an intravenous (IV) adenosine triphosphate (ATP) competitive, highly selective and potent inhibitor of pan-class I isoform phosphatidylinositol-4,5-bisphosphate 3-kinase (PI3-K) and mammalian target of rapamycin (mTOR) (Fry et al. 2004). Preclinical and first-in-human studies have shown a manageable safety profile with predictable toxicity for this class of drugs.

Activation of the PI3-K/Akt/mTOR/p-S6 pathway has been associated with endocrine resistance in ER+ breast cancer. There is ample evidence that inhibition of this pathway, in combination with anti-hormonal therapy, increases PFS (Baselga et al. 2012). There is also clinical evidence that combination therapy targeting all three pathways is feasible, safe and effective (Sweeney et al. 2014). The advantage of Gedatolisib is its potential to inhibit signaling through different PI3-K isoforms. Also important is the fact that once a week administration may be as effective, but less toxic, than chronic oral dosing. If hyperglycemia is a surrogate for effective PI3-K/Akt/mTOR/p-S6 inhibition, once weekly dosing of Gedatolisib would appear to accomplish equivalent degrees of hyperglycemia as chronically oral dosing and with less toxicity.

Preoperative or neoadjuvant systemic chemotherapy, once reserved for patients with locally advanced breast cancer in whom the goal was to render large breast cancers operable, has become increasingly common due to the improvement in disease-free survival and overall survival. Historically, the endpoint of pathological Complete Response (pCR) in neoadjuvant therapy against ER+/HER2- breast cancer has been of limited value. However, new targeted agents, with higher response rates, have the potential to use pCR assessment as a strong clinical endpoint in drug development. Given the systemic response rate in previously treated Stage 4 breast cancer patients, the expectation will be a similar high rate of pathological improvement which can lead to greater use of targeted agents in the neoadjuvant setting.

In addition to the potential of better pathological improvement, the advantage of clinical studies involving neoadjuvant therapy is that they can provide response information in patients that are treatment-naïve. This type of clinical trial can also be used to assess cellular and molecular changes with serial biopsies while on neoadjuvant therapy, which can aid in development of companion tissue and/or imaging biomarkers, and further the development of preclinical models.

Accordingly, this investigation assesses the safety and efficacy of the combination of Gedatolisib, palbociclib and faslodex in the neoadjuvant setting in previously untreated patients with ER+/HER2- breast cancer. Being the first clinical trial using this combination in neoadjuvant setting, one of the main objectives for the current trial is to determine the Maximum Tolerated Dose (MTD) of Gedatolisib when used in combination with palbociclib and faslodex. Subsequent Phase II clinical trials will be conducted to assess the safety and efficacy of the Gedatolisib/palbociclib/faslodex combination, with the dose of Gedatolisib being the MTD determined from the current trial.

ELIGIBILITY:
Inclusion Criteria:

A. Stage I-IV, with primary cancer in place, non-inflammatory invasive breast cancer confirmed by core needle or incisional biopsy (excisional biopsy is not allowed):

* the disease is ER+ (defined as ER expression >10% of invasive cancer cells according to immunohistochemical [IHC] staining)
* HER2- (defined as IHC staining of 0 to 1+ or fluorescence in situ hybridization [FISH] ratio of HER2 gene copy/chromosome 17 of <2.0.)
* the disease is previously untreated for breast cancer, operable and intend to undergo surgery for her disease (e.g., a mastectomy or lumpectomy) after completion of neoadjuvant therapy
* the disease must be measurable, defined as clinically or radiographically measureable target lesion in the breast that is ≥1 cm in diameter
* the disease cannot be axillary disease only (i.e., no identifiable tumor in the breast that is ≥1 cm on physical exam or radiographic study)
* the disease can be multi-centric or bilateral disease, provided the target lesion meets the above eligibility criteria
* breast cancer patients with lobular and luminal histology will be included. However, patients with lobular histology should not be more than a quarter of the total number of patients in this trial, as the investigational drugs are likely to have greater activities in patients with luminal histology.

(Note 1: In patients with Stage III disease, imaging studies is performed to rule out overt metastatic disease. In patients with clinically positive axillae, histologic confirmation by biopsy or fine-needle aspiration is performed. Patients with clinically negative axillae can undergo pretreatment sentinel lymph node sampling.) (Note 2: In patients with Stage IV disease, the disease must be of low burden. Low burden is defined in this study as no more than one metastatic site in the liver or lung, or up to three metastatic sites in the bone, regardless of the number of lymph nodes per latest radiographic scan. If a patient is found to have metastatic disease on scan(s) performed after patient completes study neoadjuvant therapy, surgery will not be performed and patients will be excluded from this study.)

B. Females ≥18 years of age.

C. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use effective contraceptive methods (such as abstinence, intrauterine device [IUD], or double barrier device) during the study, and must have a negative serum or urine pregnancy test within one week prior to treatment initiation.

D.Mentally competent, able to understand and willingness to sign the informed consent form.

E.At least 4 weeks must have elapsed from any prior major surgery or hormonal therapy. The following procedures are not considered major surgical procedure:

* Obtaining the required research needle biopsies
* Placement of a radiopaque clip to localize a tumor or tumors for subsequent surgical resection
* Placement of a port for central venous access
* Fine needle aspiration of a prominent or suspicious axillary lymph node
* Needle biopsy of a clinically or radiographically detected lesion to rule out metastatic diseaseF.Laboratory values ≤2 weeks must be:
* Sampling of sentinel lymph node.

F.Laboratory values ≤2 weeks must be:

* Adequate glycemic balance (hemoglobin A1c or glycated hemoglobin ≤8%; fasting serum glucose 130 mg/dL, and fasting triglycerides 300 mg/dL).
* Adequate hematology (white blood cell [WBC] 3500 cells/mm3 or 3.5 bil/L; Granulocytes ≥ 1,000/μL; platelet count 100,000 cells/mm3 or 100 bil/L; absolute neutrophil count [ANC] ≥1500 cells/mm3 or 1.5 bil/L; and hemoglobin (Hgb) ≥9 g/dL or ≥90 g/L).
* Adequate hepatic function (aspartate aminotransferase [AST/SGOT] 3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] 3x UNL (≤5x UNL if liver metastases present), bilirubin 1.5x UNL).
* Adequate renal function (serum creatinine 1.5 mg/dL or 133 µmol/L).
* Adequate coagulation (International Normalized Ratio [INR] must be <1.5, <2.3 if patient is on stable, therapeutic doses of warfarin and has no active bleeding or pathologic condition that is associated with a high risk of bleeding)

Exclusion Criteria

A.Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, symptomatic coronary artery disease, myocardial infarction within the past 6 months, uncontrolled or symptomatic cardiac arrhythmia, or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity.

B. A marked baseline prolongation of QT/QTc interval (e.g., repeated exhibition of a QTc interval >470 ms).

C. A history of additional risk factors for torsade de pointes (e.g., clinically significant heart failure, hypokalemia, family history of Long QT Syndrome).

D. Arterial thrombotic event, stroke, or transient ischemia attack within the past 12 months.

E. Uncontrolled hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure >90 mm Hg), or peripheral vascular disease ≥grade 2.

F.Active central nervous system (CNS), epidural tumor or metastasis, or brain metastasis.

G.Any active uncontrolled bleeding, a bleeding diathesis (e.g., active peptic ulcer disease), or a history of bleeding (e.g., hemoptysis, upper or lower gastrointestinal bleeding) within the past 6 months.

H.Dyspnea with minimal to moderate exertion. Patients with large and recurrent pleural or peritoneal effusions requiring frequent drainage (e.g. weekly). Patients with any amount of clinically significant pericardial effusion.

I.Diabetes of any type, except non-insulin dependent diabetes mellitus .(NIDDM) that is controlled and with hemoglobin A1c <8%.

J.Evidence of active infection during screening, or serious infection within the past month.

K.Patients with known HIV infection.

L.Serious or non-healing wound, skin ulcer, or bone fracture.

M.Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months.

N.Neuropathy of grade ≥2.

O.Albumin <2.5 g/dL or <25 g/L.

P.Lactating females.

Q.Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.

R.Unwilling or unable to follow protocol requirements.

S.Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 3 weeks prior to participating in the study.

T.Requirement for immediate palliative treatment of any kind including surgery and radiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12-24 months
  safety, tolerability,potential efficacy and MTD of Gedatolisib and MTD used in combination with palbociclib and Faslodex, in patients with

SECONDARY OUTCOMES:
Number of participants with treatment-related pathological Complete Response (pCR) | 1 year
  pCR induced by the Gedatolisib/palbociclib/Faslodex combination in the neoadjuvant setting in previously untreated patients with ER+/HER2- breast cancer. pCR assessments are performed on tissue from tumor excision surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hoffman, MD, Principal Investigator — Hoffman Oncology
Locations (2):
- United States (2):
  - California Research Institute, Los Angeles, California
  - Hoffman Oncology, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT02626507/Prot_000.pdf
  • Informed Consent Form (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT02626507/ICF_001.pdf